CLINICAL TRIAL: NCT04661410
Title: Reward Re-Training: A New Treatment to Address Reward Imbalance During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009008088; R01MH122392-01S1 (NIH)
Record Dates: First submitted 2020-12-07; First posted 2020-12-10 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bulimia Nervosa; Bulimia; Atypical; Binge Eating; Binge-Eating Disorder
Keywords: Eating Disorders; Bulimia Nervosa; Binge Eating Disorder; Binge Eating; Reward Re-training; Supportive Psychotherapy
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reward Re-Training (Experimental): 10 weekly sessions of Reward Re-Training Group Therapy.
  Interventions: Behavioral: Reward Re-Training
- Supportive Therapy (Active Comparator): 10 weekly sessions of Supportive Group Therapy.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Reward Re-Training — A brief, 10-session group-based behavioral treatment that is designed to indirectly change binge eating by directly focusing on building a more rewarding life. RRT hypothesizes that reductions in binge eating will occur as life becomes more rewarding because individuals will no longer need to rely on binge eating as a primary source of momentary reward. RRT notes that in order to live a satisfying life, individuals need to experience an adequate amount of reward in two overlapping yet distinguishable domains: momentary reward (i.e., the active experience of pleasure in the moment) and sustained reward (i.e., a deeper and more long-lasting sense of fulfillment and meaning that arises from building a personally valued life). A key aspect of RRT is an emphasize on building lasting and meaningful social relationships given the clear evidence that social connectedness can enhance both momentary reward and sustained reward.
  Arms: Reward Re-Training
Behavioral: Supportive Therapy — A brief, 10-session group-based treatment that is designed to instill hope and optimism and to increase social connection and support through a non-directive group leader that allows the patients to determine the focus of each session. The group leader will act as an empathetic provider by using reflective listening, eliciting and validating affect, and offering empathic comments.
  Arms: Supportive Therapy

SUMMARY:
In the current study, the investigators will revise our existing 10-session group RRT treatment manual to specifically address the challenges in building social support and enhancing both momentary and sustained reward during the COVID-19 pandemic (Preliminary Aim 1). In months 2-18, the investigators will conduct a small pilot RCT that will randomize individuals to receive either 10-sessions of RRT (n=30) or supportive therapy (n=30), both delivered as group-treatments via videoconferencing software. The specific aims of the current study are to confirm the feasibility and acceptability of RRT for EDs (Primary Aim 1), evaluate the ability of RRT to engage critical targets including reward to day-to-day life activities, reward to palatable foods, social isolation, and loneliness (Primary Aim 2), and provide preliminary estimates of efficacy in reducing ED symptoms at both post-treatment and a 3-month follow-up (Primary Aim 3). the investigators will also evaluate the impact of RRT on secondary outcome variables including depression, substance use, and quality of life (Secondary Aim 1).

ELIGIBILITY:
Inclusion Criteria:

1. Have experienced 12 or more loss of control episodes within the previous 3 months
2. Have a BMI above 18.5
3. Are located in the US and willing/able to participate in remote treatment and assessments
4. Are able to give consent

Exclusion Criteria:

1. Are unable to fluently speak, write and read English
2. Have a BMI below 18.5
3. Are receiving treatment for an eating disorder
4. Require immediate treatment for medical complications as a result of eating disorder symptoms
5. Have a mental handicap, or are experiencing other severe psychopathology that would limit the participants' ability to comply with the demands of the current study (e.g. severe depression with suicidal intent, active psychotic disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Stratton Hall, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] LaFata EM, Worwag K, Derrigo K, Hessler C, Allison KC, Juarascio AS, Gearhardt AN. Development of the Food Addiction Symptom Inventory: The first clinical interview to assess ultra-processed food addiction. Psychol Assess. 2024 Nov;36(11):654-664. doi: 10.1037/pas0001340. Epub 2024 Aug 5. PMID 39101915
- [Derived] Juarascio AS, Michael ML, Srivastava P, Manasse SM, Drexler S, Felonis CR. The Reward Re-Training protocol: A novel intervention approach designed to alter the reward imbalance contributing to binge eating during COVID-19. Int J Eat Disord. 2021 Jul;54(7):1316-1322. doi: 10.1002/eat.23528. Epub 2021 Apr 28. PMID 33908655

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reward Re-Training | Supportive Therapy
Started | 29 | 30
Completed | 24 | 22
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reward Re-Training | Supportive Therapy | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.79 (13.30) | 40.37 (12.36) | 40.58 (12.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Male | 5 | 7 | 12
  Sex at Birth: Female | 24 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 13 | 19 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Baseline EDE Global Score [Mean (Standard Deviation); unit: Scores on a scale] — The Eating Disorder Examination (EDE) is a diagnostic interview for the assessment of eating disorder symptoms, including binge eating frequency, compensatory behavior frequency, and global eating pathology. The EDE yields a global score and four subscale scores (Restraint, Eating concern, Shape concern, Weight concern), with higher scores indicating greater severity of eating disorder pathology. To obtain the global score, the subscale scores (which range from 0 to 6) are summed, and the resulting total is divided by the number of subscales (i.e. four).
  Scores on a scale | 2.72 (0.91) | 2.70 (0.99) | 2.71 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Frequency Assessed by the Eating Disorder Examination
Description: Frequency (number of instances) of binge eating over the past 28 days assessed by the Eating Disorder Examination
Time Frame: Each assessment time point throughout treatment (Pretreatment (Baseline), Mid-treatment (Week 5), Posttreatment (Week 10)) and a 3-month post-treatment follow-up assessment.
Measure: Mean (Standard Deviation); unit: Binge eating episodes
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
Binge eating episodes
  Binge Eating Frequency at Pretreatment | 25.10 (22.56) | 25.27 (19.09)
  Binge Eating Frequency at Mid-treatment | 9.19 (13.95) | 13.07 (15.25)
  Binge Eating Frequency at Posttreatment | 8.94 (12.10) | 8.17 (8.67)
  Binge Eating Frequency at 3-month Follow-up | 6.38 (16.77) | 4.35 (6.54)

2. Primary Outcome: Global Eating Pathology
Description: The Eating Disorder Examination is a semi-structured interview that measures eating. pathology. The EDE yields a total eating pathology score that will be used as an outcome variable. Global eating pathology is on a 0-6 point scale with higher scores indicating more significant eating pathology.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
score on a scale
  EDE Global Score at Prettreatment | 2.72 (0.91) | 2.70 (0.99)
  EDE Global Score at Mid-treatment | 2.21 (0.96) | 2.10 (0.96)
  EDE Global Score at Posttreatment | 1.87 (0.89) | 1.98 (0.78)
  EDE Global Score at 3-month Follow-up | 1.43 (0.93) | 2.04 (0.95)

3. Primary Outcome: Remission Status
Description: A participant is considered to be in remission if they had no loss of control eating episodes or compensatory behaviors in the past 28 days, as well as an EDE global score less than 1.74 (which is within one standard deviation of community norms).
Time Frame: Each assessment time point after treatment completion (Posttreatment (Week 10) and a 3-month post-treatment follow-up assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
Participants
  Remission at Posstreatment | 4 | 1
  Remission at 3-month follow-up | 7 | 6

4. Primary Outcome: Compensatory Behavior Frequency Assessed by the Eating Disorder Examination (EDE)
Description: Frequency ( number of instances) of compensatory behaviors assessed by the Eating Disorder Examination
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Compensatory behavior episodes
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
Compensatory behavior episodes
  Compensatory Behavior Frequency at Pretreatment | 5.62 (7.60) | 6.20 (12.03)
  Compensatory Behavior Frequency at Mid-treatment | 4.10 (6.83) | 4.02 (7.57)
  Compensatory Behavior Frequency at Posttreatment | 2.52 (5.60) | 2.87 (7.78)
  Compensatory Behavior Frequency at 3-month Follow-up | 1.91 (5.28) | 3.35 (8.26)

5. Secondary Outcome: Depressive Symptoms as Assessed by the Beck Depression Inventory-II
Description: Assesses the type (description of certain feelings or attitudes) and intensity (how often or how much the feelings and attitudes are present) of various depressive symptoms using a total score. The scale ranges from 0-63 with higher scores indicating worse depressive symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
Score on a scale
  BDI Score at Pretreatment | 15.83 (11.10) | 18.87 (10.38)
  BDI Score at Mid-treatment | 10.19 (10.87) | 14.95 (8.75)
  BDI Score at Posttreatment | 9.57 (10.70) | 13.30 (10.89)
  BDI Score at 3-month Follow-up | 7.94 (9.32) | 17.02 (4.51)

6. Secondary Outcome: Substance Use Assessed by the NIDA-Modified ASSIST
Description: Frequency of substance use (number of days/month) assessed by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
days/month
  Frequency of Substance Use at Pretreatment | 3.00 (4.70) | 2.83 (4.00)
  Frequency of Substance Use at Mid-treatment | 3.31 (4.95) | 2.50 (3.70)
  Frequency of Substance Use at Posttreatment | 2.93 (6.29) | 2.03 (3.70)
  Frequency of Substance Use at 3-month Follow-up | 2.90 (5.64) | 2.57 (4.57)

7. Secondary Outcome: Quality of Life Assessed by the Quality of Life Inventory (QOLI)
Description: Assesses the importance of 16 given life domains have on influencing happiness and current satisfaction level regarding these 16 life domains. Scores range from 1-77 with higher scores indicating better quality of life.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Reward Re-Training | Supportive Therapy
Number analyzed (Participants) | 29 | 30
Score on a scale
  QOLI Scores at Pretreatment | 15.48 (1.96) | 15.59 (2.11)
  QOLI Scores at Mid-Treatment | 16.04 (1.50) | 15.92 (2.04)
  QOLI Scores at Posttreatment | 16.33 (1.60) | 16.32 (1.89)
  QOLI Scores at 3-month Follow-up | 16.16 (1.84) | 16.22 (1.99)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Reward Re-Training | Supportive Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04661410/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04661410/SAP_001.pdf